CLINICAL TRIAL: NCT04916327
Title: Examining the Impact of Exercise Training on Vascular Dysfunction in Individuals With Mental Health Disorders - Study 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HM20020955-1
Record Dates: First submitted 2021-05-24; First posted 2021-06-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Vascular Diseases
Keywords: cardiovascular disease; vascular function; PTSD; GAD; Oxidant
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases; Stress Disorders, Post-Traumatic | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant then Placebo (Experimental): Subjects will ingest an antioxidant cocktail prior to their second visit and a placebo prior to third second visit
  Interventions: Dietary Supplement: Antioxidant; Dietary Supplement: Placebo
- Placebo then Antioxidant (Experimental): Subjects will ingest a placebo prior to their second visit and an antioxidant cocktail prior to their third visit.
  Interventions: Dietary Supplement: Antioxidant; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidant — Subjects will ingest an antioxidant cocktail containing 800 milligrams of alpha lipoic acid, 1 gram of vitamin C (ascorbic acid), and 400 milligrams of vitamin E (alpha tocopherol).
Dietary Supplement: Placebo — Subjects will ingest placebo (microcrystalline cellulose) pills.

SUMMARY:
The purpose of this research study is to examine the role oxidants, substances produced in the blood that can damage blood vessel function, may play in blood vessel function in healthy individuals as well as individuals with mental health disorders (posttraumatic stress disorder (PTSD) and/or generalized anxiety disorder (GAD)).

DETAILED DESCRIPTION:
Study #1 is made up of three sessions done on three separate days and the entire study can be completed in as little as two weeks. All testing sessions will take place at the Exercise Physiology Research Laboratory. Volunteers will be asked to participate in one initial testing session (Visit 1) lasting < 1 hour that will help make them more familiar with the study equipment and procedures, determine body measures (height, weight, body fat), determine the maximum strength of their forearm and calf, and require one blood draw. The following two testing sessions (Visits 2 and 3) with each session lasting between 2-3 hours that will involve multiple tests designed to determine the health of their blood vessels. For Visit #2 they will be randomly given either antioxidant pills or placebo pills to determine the effect of oxidants on blood vessel health. For Visit #3, they will be given whatever set of pills (antioxidant or placebo) that they did not receive during Visit #2.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy and free of overt cardiovascular, pulmonary, or metabolic disease
* for PTSD group, a score of ≥ 33 on PCL-5 checklist
* for GAD group, a score of ≥ 10 on the GAD-7 self-report scale and < 33 on the PCL-5 checklist
* for Healthy Control group, a score of ≤ 10 on the GAD-7 self-report scale and < 33 on the PCL-5 checklist

Exclusion Criteria:

* taking medications that could influence cardiovascular function
* current smokers who have recently quit smoking
* illicit drug use or excessive alcohol consumption
* pregnant women
* significant calorie restriction or vitamin/mineral deficiencies
* limited English proficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 720 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Arm Vascular Function at Rest (Flow Mediated Dilation Test) | Baseline to the end of the final visit, about 2 weeks
  Change in Brachial Artery Dilation from Baseline Values
Leg Vascular Function (Passive Leg Movement Test) | Baseline to the end of the final visit, about 2 weeks
  Change in Leg Blood Flow Values from Baseline
Arm Vascular Function in Response to Exercise (Handgrip Exercise Test) | Baseline to the end of the final visit, about 2 weeks
  Change in Brachial Artery Dilation from Baseline Values

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Garten, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States